CLINICAL TRIAL: NCT02897440
Title: Full Repairing Versus Partial Repairing of Soft Tissue Surrounding the Hip Joint in Hip Arthroplasty for Femoral Neck Fractures
Brief Title: Full Versus Partial Repairing of Soft Tissue Surrounding the Hip in Arthroplasty for Femoral Neck Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Hospitals affiliated to the China PLA General Hospital (Other Government)
Responsible Party: Principal Investigator, Haibo Lu, Attending Surgeon, First Hospitals affiliated to the China PLA General Hospital
Other Study IDs: 1
Record Dates: First submitted 2016-08-24; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Femoral Neck Fracture
Keywords: Femoral Neck Fracture; Hip Arthroplasty; Repairing of soft tissue
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Full Repairing of soft tissue surrounding the hip: Full repairing soft tissue surrounding the hip damaged during the procedure of hip dislocation and prosthesis implanting
  Interventions: Procedure: Full Repairng of soft tissue surrounding the hip
- Partial Repairing of soft tissue surrounding the hip: Partial repairing soft tissue surrounding the hip damaged during the procedure of hip dislocation and prosthesis implanting
  Interventions: Procedure: Partial Repairng of soft tissue surrounding the hip

INTERVENTIONS:
Procedure: Full Repairng of soft tissue surrounding the hip — Full repairing soft tissue surrounding the hip damaged during the procedure of hip dislocation and prosthesis implanting.
  Groups: Full Repairing of soft tissue surrounding the hip
Procedure: Partial Repairng of soft tissue surrounding the hip — Partial repairing soft tissue surrounding the hip damaged during the procedure of hip dislocation and prosthesis implanting.
  Groups: Partial Repairing of soft tissue surrounding the hip

SUMMARY:
A prospective cohort study to compare full repairing and partial repairing of soft tissue surrounding the hip joint in anteriorolateral approaching arthroplasty concerning hip function. Patients admitted with a femoral neck fracture operated with a hip arthroplasty through an anteriorolateral approach were screened for inclusion. Patients with altered mental status SPMSQ <7, pathological fractures, non-walkers were excluded.

DETAILED DESCRIPTION:
Those who fulfilled the inclusion criteria and non of the exclusion criteria were followed 2 months postoperatively by clinical examination. Sample size were estimated to 15 patients in each group. Primary outcome variables were trendelenburg test, abductor strength measured with dynamometry. Secondary outcome variables were WOMAC, EQ-5D, and VAS scores.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Walker
* Hemiarthroplasty or Total Hip Arthroplasty
* Preiffer test >7/10

Exclusion Criteria:

* Pathological fracture
* Non-walker
* Pfeiffer test <7/10 indicating mental alteration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with femoral neck fractures undergoing hip arthroplasty through anteriorolateral approach.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Trendelenburg Test | At 4 week postoperatively
  30 seconds standing on the operated leg
Abductor strength | At 4 week postoperatively
  Dynamometry

SECONDARY OUTCOMES:
WOMAC | At 2, 4, 6 weeks and 12 months postoperatively
  An established hip score
Quality of life (EQ-5D) | At 2, 4, 6 weeks and 12 months postoperatively
  EQ-5D
Pain (Visual analouge scale) | At 2, 4, 6 weeks and 12 months postoperatively
  Visual analouge scale (VAS): At rest and during activity

IPD SHARING:
Plan to Share IPD: No